CLINICAL TRIAL: NCT05896631
Title: The Effect of Spinal Anesthesia Methods on Hemodynamics in Geriatric Patients
Brief Title: The Effect of Spinal Anesthesia on Hemodynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Fatma Kavak Akelma, Anesthesiology and reanimation assistant doktor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: geriatrics
Record Dates: First submitted 2023-05-22; First posted 2023-06-09 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia, Spinal
Keywords: hemodynamic management; spinal anesthesia; geriatric anesthesia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7.5 mg hyperbaric bupivacaine (Active Comparator): Patients undergoing spinal anesthesia in the lateral decubitus position with 7.5 mg of hyperbaric bupivacaine will be included.
  Interventions: Other: 7.5 mg hyperbaric bupivacaine
- 5 mg hyperbaric bupivacaine (Active Comparator): Patients undergoing spinal anesthesia in the lateral decubitus position with 5 mg of hyperbaric bupivacaine will be included.
  Interventions: Other: 5 mg hyperbaric bupivacaine

INTERVENTIONS:
Other: 7.5 mg hyperbaric bupivacaine — Spinal anesthesia with 7.5 mg hyperbaric bupivacaine after preoperative peng (pericapsular nerve group) block
  Arms: 7.5 mg hyperbaric bupivacaine
Other: 5 mg hyperbaric bupivacaine — Spinal anesthesia with 5 mg hyperbaric bupivacaine after preoperative peng (pericapsular nerve group) block
  Arms: 5 mg hyperbaric bupivacaine

SUMMARY:
In this study, it was planned to provide more stable hemodynamics in geriatric patients with low-dose spinal anesthesia. We will compare 7.5mg hyperbaric bupivacaine with 5mg hyperbaric bupivacaine.

The researchers hypothesized that low-dose bupivacaine would provide adequate anesthesia, less hypotension, and faster recovery.

DETAILED DESCRIPTION:
Hypothesis It is hypothesized that low-dose bupivacaine can provide adequate anesthesia, less hypotension, and faster recovery.

patient population Patients over 65 years of age who will undergo spinal anesthesia due to hip fracture.

Hemodynamic data(Blood pressure-mmHg, heart rate-beats per minute) of patients, bromage scores, perfusion index (PI) values, discharge time, pain with NRS (numerical rating scale), patient satisfaction will be evaluated ( Numeric output from 1-10).

Hemodynamic variables will be recorded every 2 minutes in the first 20 minutes after spinal anesthesia. hemodynamic variables will be recorded 30 minutes after spinal anesthesia and at the end of the operation.

The perfusion index is the ratio of the blood volume to the pulsatile to non-pulsatile fraction. An increase in the pulsatile fraction that occurs during vasodilation corresponds to a higher PI. Therefore, patients with a higher PI have a higher risk of post-spinal hypotension.

ELIGIBILITY:
Inclusion Criteria:

* ASA(American Society of Anesthesiologists) I-II-III patients
* BMI( body mass index) in the range of 18-40
* over 65 years old hip fracture

Exclusion Criteria:

* Refusal to participate in the study
* Left ventricular ejection fraction below 40%
* cardiac arrhythmia
* Patients with peripheral vascular disease
* Failure of spinal anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
hemodynamic variability | every 2 minutes for the first 20 minutes after spinal anesthesia
  intraoperative hemodynamic variables (BP(blood pressure-mmHg) during hip surgery
hemodynamic variability | at 30 minutes of spinal anesthesia
  intraoperative hemodynamic variables (BP(blood pressure-mmHg) during hip surgery

SECONDARY OUTCOMES:
perfusion index variability | every 2 minutes for the first 20 minutes after spinal anesthesia
  To correlate between perfusion index and hypotension after spinal anaesthesia in hip surgery
perfusion index variability | at 30 minutes of spinal anesthesia
  To correlate between perfusion index and hypotension after spinal anaesthesia in hip surgery
perfusion index variability | at the end of the operation
  To correlate between perfusion index and hypotension after spinal anaesthesia in hip surgery
Sensory Levels | 24 hours
  Sensory levels will be measured every 30 minutes until discharge from PACU(post-anaesthesia care unit)
ephedrine use | 24 hours
  ephedrine consumption , mg in hip surgery
fentanyl use | 24 hours
  fentanyl consumption , mcg in hip surgery
bromage scale | 24 hours
  Bromage Scores every 30 minutes until discharge from PACU(post-anaesthesia care unit).
NRS(numerical rating scale) | 2 hours
  pain scoring a score of 1 to 10
NRS(numerical rating scale) | 8 hours
  pain scoring a score of 1 to 10
NRS(numerical rating scale) | 16 hours
  pain scoring a score of 1 to 10
NRS(numerical rating scale) | 24 hours
  pain scoring a score of 1 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No